CLINICAL TRIAL: NCT03621748
Title: Randomized Control Trial for Awake vs. Asleep Craniotomy for Non-eloquent Gliomas
Brief Title: Awake vs. Asleep Craniotomy for Non-eloquent Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kaisorn L. Chaichana, Senior Associate Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-005248
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Intracranial Glioma
Keywords: craniotomy; awake craniotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Awake Cohort (Active Comparator): Cohort undergoing craniotomy utilizing general anesthesia protocol
  Interventions: Procedure: Non-awake Anesthesia Protocol
- Awake Cohort (Experimental): Cohort undergoing craniotomy utilizing awake anesthesia protocol
  Interventions: Procedure: Awake Anesthesia Protocol

INTERVENTIONS:
Procedure: Awake Anesthesia Protocol — Awake is defined as the patient being awake with electrical brain stimulation mapping during the critical portions of the procedure.
  Arms: Awake Cohort
Procedure: Non-awake Anesthesia Protocol — Non-awake is general anesthesia as per convention with intubation.
  Arms: Non-Awake Cohort

SUMMARY:
This study protocol examines a comparison between local and general anesthesia (Awake vs. Asleep Craniotomy) in the removal of brain tumors that are in areas of the brain that do not directly control bodily functions (non-eloquent gliomas).

DETAILED DESCRIPTION:
This is a single-center, prospective randomized open or non-blinded end-point (PROBE) clinical trial. Patients will be selected by the neurosurgeon according to the inclusion and exclusion criteria. Patients who consent to randomization will have confirmed non-eloquent status confirmed by independent surgeon and will be randomized into 1 of 2 treatment groups utilizing a dynamic minimization approach. The experimental group with randomization of patients who will undergo awake craniotomy for both high and low grade gliomas in non-eloquent areas or a control group of patients who will have asleep craniotomy for both high and low grade gliomas in non-eloquent regions.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients with age ≥18 years old.
2. WHO grade I, II, III, and IV Glioma in non-eloquent brain cortex based on magnetic resonance imaging (MRI)
3. An elective procedure.
4. A single lesion.
5. No major comorbidities that would necessitate an extended hospital stay.
6. Newly diagnosed tumors.

EXCLUSION CRITERIA

1. Patients with age < 18 years old.
2. Non-gliomas
3. Eloquent location (motor, sensory, language)
4. Non-elective procedure.
5. Multiple lesions.
6. Major comorbidities.
7. Recurrent tumors.
8. Patients lacking capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Extent of resection | up to 48 hrs post operation
  Extent of resection (EOR) defined as the residual volume, in cm3, of tumor measured by MRI

SECONDARY OUTCOMES:
Percentage of baseline tumor volume resected | up to 48 hrs post operation
  Measured by MRI
VAS Postoperative anxiety | Day 1(+14 days) , Post op day 0, 1, 2 weeks, 3mth
  Postoperative Anxiety scale measured using a 0 to 10 visual analog scale (0: no anxiety, 10: worst anxiety)
Length of Surgery | Intraoperative
  defined as time entering OR and leaving OR

OTHER OUTCOMES:
Length of hospital stay (LOS) | 0-30 days post operation
  admission to discharge
The Karnofsky Performance Score | Day 1 (+14 days), Post-operative up to 48 hrs, 3-6 weeks, 3mths, 6mths, and 9 mths
  (KPS) ranking runs from 100 to 0, where 100 is "perfect" health and 0 is death
FACT-Br | Day 1 (+14 days), Post-operative up to 48 hrs, 3-6 weeks, 3mths, 6mths, and 9 mths
  The FACT-Brain (FACT-Br) provides an additional set of disease-specific questions pertaining to brain neoplasms
Post-operative pain scale | Day 1 (+14 days), Post-operative up to 48 hrs, 3-6 weeks, 3mths, 6mths, and 9 mths
  0 to 10 (0: No pain, 10: Worst pain) - Numeric Scale
Cost of treatment | captured until 30 days post operation
  Analysis to include standardized cost, physician service cost, cost of hospitalization and 30 days post-hospitalization cost

CONTACTS AND LOCATIONS:
Overall Officials: Kaisorn L Chaichana, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials